CLINICAL TRIAL: NCT03902951
Title: A Single-Arm, Open-Label, Phase II Study of Systemic and Tumor Directed Therapy for Recurrent Oligometastatic M1 Prostate Cancer
Brief Title: Antiandrogen Therapy and SBRT in Treating Patients With Recurrent, Metastatic Prostate Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: Janssen Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-001037; NCI-2019-00337 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2019-04-03; First posted 2019-04-04 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Metastatic Prostate Adenocarcinoma; Prostate Adenocarcinoma With Focal Neuroendocrine Differentiation; Recurrent Prostate Carcinoma; Stage IVB Prostate Cancer AJCC v8
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Abiraterone Acetate; apalutamide; Leuprolide; luprolide acetate gel depot; Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Treatment (leuprolide, apalutamide, abiraterone acetate, SBRT) (Experimental): Patients receive leuprolide SC on day 1, Patients receive a single dose of leuprolide SC on day 1 and apalutamide PO QD and abiraterone acetate PO QD for up to 6 months in the absence of disease progression or unacceptable toxicity. Beginning 2 months of initiation of ADT, patients also receive SBRT over 1, 3, or 5 fractions in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Abiraterone Acetate; Drug: Apalutamide; Drug: Leuprolide Acetate; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Radiation: Stereotactic Body Radiation Therapy

INTERVENTIONS:
Drug: Abiraterone Acetate — Given PO
  Other Names: CB7630; Zytiga
Drug: Apalutamide — Given PO
  Other Names: ARN 509; ARN-509; ARN509; JNJ 56021927; JNJ-56021927
Drug: Leuprolide Acetate — Given SC
  Other Names: A-43818; Abbott 43818; Abbott-43818; Carcinil; Depo-Eligard; Eligard; Enanton; Enantone; Enantone-Gyn; Ginecrin; LEUP; Leuplin; Leuprorelin Acetate; Lucrin; Lucrin Depot; Lupron; Lupron Depot; Lupron Depot-3 Month; Lupron Depot-4 Month; Lupron Depot-Ped; Procren; Procrin; Prostap; TAP-144; Trenantone; Uno-Enantone; Viadur
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies
Radiation: Stereotactic Body Radiation Therapy — Undergo SBRT
  Other Names: SABR; SBRT; Stereotactic Ablative Body Radiation Therapy

SUMMARY:
This phase II trial studies how well antiandrogen therapy (leuprolide, apalutamide, and abiraterone acetate) and stereotactic body radiation therapy (SBRT) works in treating patients with prostate cancer that has come back and has spread to other parts of the body. Drugs used in chemotherapy, such as leuprolide, apalutamide, and abiraterone acetate, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. SBRT uses special equipment to position a patient and deliver radiation to tumors with high precision. This method can kill tumor cells with fewer doses over a shorter period and cause less damage to normal tissue. Giving antiandrogen therapy and SBRT may work better in treating patients with prostate cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the efficacy of combined systemic and tumor directed therapy for recurrent oligometastatic M1a,b prostate cancer patients with 1-5 metastases (exclusive of pelvic nodal N1 metastases) staged by prostate-specific membrane antigen (PSMA) positron emission tomography (PET)-computed tomography (CT).

SECONDARY OBJECTIVES:

I. Time to biochemical progression. II. Time to additional antineoplastic therapy. III. Prostate cancer specific survival. IV. Safety and tolerability. V. Assessment of health related quality of life using the Functional Assessment of Cancer Therapy - Prostate (FACT-P) scale.

CORRELATIVE OBJECTIVES:

I. To determine genomic and transcriptomic features present in metastatic tumors in patients that respond to this multimodal therapy.

II. To evaluate biomarkers of response using circulating tumor cells (CTCs). III. To evaluate biomarkers of response using circulating tumor deoxyribonucleic acid (DNA) (ctDNA).

IV. To evaluate immunophenotypes of circulating immune cells.

OUTLINE:

Patients receive a single dose of leuprolide subcutaneously (SC) on day 1 and apalutamide orally (PO) once daily (QD) and abiraterone acetate PO QD for up to 6 months in the absence of disease progression or unacceptable toxicity. Beginning 2 months of initiation of antiandrogen therapy (ADT), patients also receive SBRT over 1, 3, or 5 fractions in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up within 2 -4 weeks, every 30 days for 6 months, and then every 3 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of prostate adenocarcinoma after radical prostatectomy (primary small cell carcinoma of the prostate is not allowed, however adenocarcinoma with neuroendocrine differentiation is allowed)
* Presence of 1-5 visible metastases (by PSMA PET-CT)

  * At least one metastasis must be M1a-b
  * Visceral metastases are not allowed
  * Patients may have any number of pelvic nodal metastases (but largest must be < 2 cm)
  * Metastases must be amenable to treatment with SBRT
  * Biopsy of one metastasis must be attempted, unless unsafe to perform
* Patient must be fit to undergo SBRT to all visible sites of metastases, ADT
* Total testosterone > 150 ng/dL prior to ADT (optimal time to measure total testosterone is between 8 and 9 am)
* Adequate performance status (Eastern Cooperative Oncology Group [ECOG] 0-1)
* Hemoglobin >= 9.0 g/dL, independent of transfusion and/or growth factors within 3 months prior to randomization
* Platelet count >= 100,000 x 10^9/uL independent of transfusion and/or growth factors within 3 months prior to randomization
* Serum albumin >= 3.0 g/dL
* Glomerular filtration rate (GFR) >= 45 mL/min
* Serum potassium >= 3.5 mmol/L
* Serum total bilirubin =< 1.5 x upper limits of normal (ULN)

  * Note: In subjects with Gilbert?s syndrome, if total bilirubin is > 1.5 x ULN, measure direct and indirect bilirubin and if direct bilirubin is =< 1.5 x ULN, subject may be eligible
* Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) < 2.5 x ULN
* Medications known to lower the seizure threshold must be discontinued or substituted at least 4 weeks prior to study entry

Exclusion Criteria:

* Any evidence of spinal cord compression (radiological or clinical)
* Prior pelvic malignancy
* Prior pelvic radiation aside from salvage prostate radiation
* Concurrent malignancy aside from superficial skin cancers or superficial bladder tumors
* Inability to undergo radiotherapy, or ADT
* Primary small cell carcinoma of the prostate (prostate adenocarcinoma with neuroendocrine differentiation is allowed)
* Inflammatory bowel disease or active collagen vascular disease
* History of any of the following:

  * Seizure or known condition that may pre-dispose to seizure (e.g. prior stroke within 1 year to randomization, brain arteriovenous malformation, Schwannoma, meningioma, or other benign central nervous system [CNS] or meningeal disease which may require treatment with surgery or radiation therapy)
  * Severe or unstable angina, myocardial infarction, symptomatic congestive heart failure, arterial or venous thromboembolic events (eg, pulmonary embolism, cerebrovascular accident including transient ischemic attacks), or clinically significant ventricular arrhythmias within 6 months prior to randomization
* Current evidence of any of the following:

  * Uncontrolled hypertension
  * Gastrointestinal disorder affecting absorption
  * Active infection (eg, human immunodeficiency virus [HIV] or viral hepatitis)
  * Any chronic medical condition requiring a higher dose of corticosteroid than 10 mg prednisone/prednisolone once daily
  * Any condition that in the opinion of the investigator would preclude participation in this study
  * Concomitant strong CYP3A4 inducers. (If a strong CYP3A4 inducer must be co-administered, abiraterone acetate dose frequency will be adjusted). [SAFETY: Warning against use with CYP2C8 inhibitors with narrow therapeutic index is also pertinent to be included as it is also part of United States Prescribing Information (USPI): In a CYP2C8 drug-drug interaction trial in healthy subjects, the area under curve (AUC) of pioglitazone (CYP2C8 substrate) was increased by 46% when pioglitazone was given together with a single dose of 1,000 mg abiraterone acetate. Therefore, patients should be monitored closely for signs of toxicity related to a CYP2C8 substrate with a narrow therapeutic index if used concomitantly with ZYTIGA]
  * Treatment with CYP2D6 substrates that have a narrow therapeutic index. If an alternative treatment cannot be used, a dose reduction of the CYP2D6 substrate may be considered
  * Baseline moderate and severe hepatic impairment (ChildPugh Class B & C)
* Presence of visceral metastases (i.e., stage M1c)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2021-03-17 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Percent of patients achieving a serum prostate specific antigen (PSA) of < 0.05 ng/mL | Up to 6 months post treatment
  Will be summarized by count and percent along with the 95% confidence interval.

SECONDARY OUTCOMES:
Time to biochemical progression | Baseline to first rise in PSA to 0.2 ng/mL, assessed up to 2 years
  Will be summarized using Kaplan-Meier method.
Time to radiographic progression | Baseline to time when any imaging shows new evidence of metastatic disease, assessed up to 2 years
  Will be summarized using Kaplan-Meier method.
Time to initiation of alternative antineoplastic therapy | Baseline to time when new anti-prostate cancer therapy is initiated, assessed up to 2 years
  Will be summarized using Kaplan-Meier method.
Prostate cancer specific survival | Up to 2 years post treatment
Health related quality of life: Functional Assessment of Cancer Therapy - Prostate (FACT-P) scale - patient questionnaire | Up to 2 years post treatment
  This uses the Functional Assessment of Cancer Therapy - Prostate (FACT-P) questionnaire. It assesses patient function in four domains: Physical, Social/Family, Emotional, and Functional well-being, which is further supplemented by 12 site specific items to assess for prostate related symptoms. Items are rated on a 0 to 4 Likert type scale and combined to produce subscale scores for each domain and a global score, the higher the score, the better the quality of life. Range from 0-150 . Data will be aggregated per patient and over time.
Incidence of adverse events | Up to 30 days post treatment
  The intensity of clinical adverse events will be graded according to the Common Terminology Criteria for Adverse Events version (v) 4.0 (CTCAE) grading system in the toxicity categories.
Biomarker analysis | Up to 2 years post treatment
  Will conduct whole exome deep sequencing (WES), RNA sequencing (RNA-seq), and comparative genomic hybridizations (CGH) of the metastatic tumors.

OTHER OUTCOMES:
Genomic and transcriptomic features present in metastatic tumors | Up to 2 years post treatment
  Will conduct whole exome deep sequencing (WES), ribonucleic acid (RNA) sequencing (RNA-seq), and comparative genomic hybridizations (CGH) of the metastatic tumors of the 28 patients enrolled in the Phase II trial. Then, will identify discriminating features of the metastatic tumors in responders that distinguish them from the non-responders.
Circulating tumor deoxyribonucleic acid (ctDNA) for predictors of response | Up to 2 years post treatment
Circulating tumor cells (CTCs) for predictors of response | Up to 2 years post treatment
Changes in circulating immunophenotypes | Baseline up to 2 years post treatment

CONTACTS AND LOCATIONS:
Overall Officials: Amar Kishan, Principal Investigator — UCLA / Jonsson Comprehensive Cancer Center
Locations (1):
- UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California, United States

REFERENCES:
- [Derived] Nikitas J, Rettig M, Shen J, Reiter R, Lee A, Steinberg ML, Valle LF, Sachdeva A, Romero T, Calais J, Czernin J, Nickols NG, Kishan AU. Systemic and Tumor-directed Therapy for Oligorecurrent Metastatic Prostate Cancer (SATURN): Primary Endpoint Results from a Phase 2 Clinical Trial. Eur Urol. 2024 Jun;85(6):517-520. doi: 10.1016/j.eururo.2024.01.021. Epub 2024 Mar 16. PMID 38494380